CLINICAL TRIAL: NCT00653809
Title: Elucidating the Role of Nitric Oxide and Endothelin-1 Activation in Endothelial Cells Co-cultured With Placental Explants From African-american and Caucasian High Risk Pregnancies
Brief Title: Racial Differences: Nitric Oxide(NO) and Endothelin-1(ET-1) in Preeclampsia (PreE)
Status: Completed | Type: Observational
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Office of Minority Health (Unknown); Mississippi Institute for Improvement of Geographic Minority Health (Unknown)
Responsible Party: Principal Investigator, Kedra Wallace, Postdoc Research Fellow, University of Mississippi Medical Center
Other Study IDs: 2007-0065
Record Dates: First submitted 2008-04-01; First posted 2008-04-07 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Placental Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- A, 1, I: Caucasian women without preeclampsia or PIH, delivering their first child
- A, 1, II: Caucasian women with preeclampsia or PIH, delivering their first child
- A, 2, I: African-american women without preeclampsia or PIH, delivering their first child
- A, 2, II: African-American women with preeclampsia or PIH, delivering their first child
- B, 1, I: Caucasian women without preeclampsia or PIH, delivering at least their second child
- B, 1, II: Caucasian women with preeclampsia or PIH, delivering at least their second child
- B, 2, I: African-american women without preeclampsia or PIH, delivering at least their second child
- B, 2, II: African-american women with preeclampsia or PIH, delivering at least their second child

SUMMARY:
The goal of this study is to examine the activation of markers of endothelial and cardiovascular dysfunctions, from women with high-risk pregnancies. Information from this study will hopefully provide enough information to determine a link between race, the advent of high risk pregnancies and cardiovascular markers. With this information it might be possible to intervene with approved pharmacological treatments.

ELIGIBILITY:
Inclusion Criteria:

* African-american or Caucasian
* Pregnant
* Between ages of 18 - 40 years of age

Exclusion Criteria:

* Presence of a disease or condition which is not preeclampsia
* Drug or alcohol abuse during pregnancy
* Obesity

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women delivering babies at the University of MS Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2007-06; Primary Completion 2008-12 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Nitric oxide and Endothelin-1 levels | 48 hours after tissue collection

SECONDARY OUTCOMES:
Nitric oxide isoforms and Endothelin-1 receptor activation based on primary outcome | within 6 months from tissue collection

CONTACTS AND LOCATIONS:
Overall Officials: Kedra L Wallace, PhD, Principal Investigator — Obstetrics & Gynecology
Locations (1):
- University of MS Medical Center, Jackson, Mississippi, United States